CLINICAL TRIAL: NCT02096692
Title: ProMRI Study of the Iforia ICD System (Phase C)
Status: Completed | Type: Observational
Sponsor: Biotronik, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: G120226 (Phase C)
Record Dates: First submitted 2014-03-24; First posted 2014-03-26 (Estimated); Results first posted 2015-10-22 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-02

CONDITIONS: Implantable Cardioverter-Defibrillator With Magnetic Resonance Imaging
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- ICD System Therapy: Patients with a ProMRI ICD System
  Interventions: Device: Patients with a ProMRI ICD System; Other: Magnetic Resonance Imaging (MRI) scan

INTERVENTIONS:
Device: Patients with a ProMRI ICD System — Tachycardia Fast Heart Beat
Other: Magnetic Resonance Imaging (MRI) scan — MRI scan of heart/chest or thoracic spine

SUMMARY:
The objective of the ProMRI Study is to demonstrate the clinical safety of the ProMRI ICD System when used under specific MRI conditions.

ELIGIBILITY:
Inclusion Criteria:

The following initial inclusion criteria must be met for a subject to be enrolled and considered for the MRI-procedure:

* Age greater than or equal to 18 years
* Able and willing to complete MRI testing
* Able to provide written informed consent
* Available for follow-up visit at the study site
* Implanted with an ICD System consisting only of an Iforia DR-T and Linoxsmart S 65 / Linoxsmart SD 65/18 with Setrox S 53 atrial lead or Iforia VR-T DX and Linoxsmart S DX 65/15 or Linoxsmart S DX 65/17.
* ICD implanted pectorally
* All ICD system components implanted, repositioned, or exchanged at least 5 weeks prior to enrollment
* Underlying rhythm identifiable during sensing test
* All pacing thresholds are measureable and are less than or equal to 2.0 V @ 0.4 ms (Criterion does not apply to atrial pacing threshold for subjects with an Iforia DR-T that have AF and are permanently programmed to VVI and for subjects with an Iforia VR-T DX)
* Ventricular sensing is measurable and >6.5mV
* Absence of phrenic nerve stimulation at 5.0V and 1.0 ms
* Pacing impedance is between 200 and 1500 ohm
* Shock Impedance is between 30 and 90 ohm
* Able and willing to use the CardioMessenger II

At the pre-MRI procedure, the following procedure-related criteria must be met for the subject to undergo the MRI scan:

* Absence of phrenic nerve stimulation at 5.0V @ 1.0 ms
* |pacing threshold at Pre-MRI follow-up - pacing threshold at baseline| ≤ 0.5 V (ICD Lead Only)
* All pacing thresholds are measureable and are less than or equal to 2.0 V @ 0.4 ms (Criterion does not apply to atrial pacing threshold for subjects with an Iforia DR-T that have AF and are permanently programmed to VVI and for subjects with an Iforia VR-T DX.)
* Ventricular sensing is measurable and >6.5mV
* The ICD system has been implanted for at least six weeks.
* Subject did not have an ICD or lead explant, exchange or reposition in the previous 6 weeks.
* All lead pacing impedances are between 200 and 1500 ohm
* Shock impedance is between 30 and 90 ohm
* Battery status is at least 30% of capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients selected for participation should be from the investigators' general patient population according to the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2014-06; Primary Completion 2015-03 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (38):
- United States (38):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Concord, California
  - Newport Beach, California
  - Rancho Mirage, California
  - New Haven, Connecticut
  - Newark, Delaware
  - Washington D.C., District of Columbia
  - Valparasio, Indiana
  - Iowa City, Iowa
  - Lafayette, Louisiana
  - Cumberland, Maryland
  - Takoma Park, Maryland
  - Boston, Massachusetts
  - Burlington, Massachusetts
  - Worcester, Massachusetts
  - Ann Arbor, Michigan
  - Grand Rapids, Michigan
  - Ypsilanti, Michigan
  - Kansas City, Missouri
  - St Louis, Missouri
  - Flushing, New York
  - New York, New York
  - The Bronx, New York
  - Winston-Salem, North Carolina
  - Columbus, Ohio
  - Toledo, Ohio
  - Portland, Oregon
  - Salem, Oregon
  - Langhorne, Pennsylvania
  - Wynnewood, Pennsylvania
  - Greenville, South Carolina
  - Nashville, Tennessee
  - Amarillo, Texas
  - Mechanicsville, Virginia
  - Virginia Beach, Virginia
  - Spokane, Washington

REFERENCES:
- [Result] Awad K, Griffin J, Crawford TC, Lane Cox S, Ferrick K, Mazur A, Pena RE, Lloyd SG, Michalski J, Johnson W, Bailey WM. Clinical safety of the Iforia implantable cardioverter-defibrillator system in patients subjected to thoracic spine and cardiac 1.5-T magnetic resonance imaging scanning conditions. Heart Rhythm. 2015 Oct;12(10):2155-61. doi: 10.1016/j.hrthm.2015.06.002. Epub 2015 Jun 3. PMID 26049048

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ICD System Therapy
Started | 154
Completed | 150
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | ICD System Therapy
Number analyzed (Participants) | 154
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 119

OUTCOME MEASURES:

1. Primary Outcome: MRI and ICD System Related Serious Adverse Device Effect (SADE) Free Rate
Time Frame: 1 Month Post-MRI
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ICD System Therapy
Number analyzed (Participants) | 154
percentage of participants | 100 [97.6 to 100]

2. Primary Outcome: Percentage of Participants Free of Ventricular Pacing Threshold Rise
Description: Evaluate the percentage of ICD leads free of ventricular pacing threshold increase between the Pre-MRI and one-month post-MRI follow-up.
Time Frame: Between Pre-MRI and 1 Month Post-MRI
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ICD System Therapy
Number analyzed (Participants) | 154
percentage of participants | 100 [97.6 to 100]

3. Primary Outcome: Percentage of Participants Free of R-wave Sensing Attenuation
Description: Evaluate the percentage of subjects free of R-wave attenuation between the Pre-MRI and one-month post-MRI follow-up.
Time Frame: Between Pre-MRI and 1 Month Post-MRI
Population: All participants who had measurable R-waves at both pre-MRI and and 1 Month Post-MRI.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ICD System Therapy
Number analyzed (Participants) | 153
percentage of participants | 99.3 [96.4 to 100]

ADVERSE EVENTS:
Arm/Group | ICD System Therapy
Serious Adverse Events (participants affected / at risk) | 23/154
Other Adverse Events (participants affected / at risk) | 24/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ICD System Therapy (N=154)
Angina (Cardiac disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 2 (2)
Cardiac Arrest (Cardiac disorders) | 1 (1)
Infection (General disorders) | 6 (6)
Influenza (Infections and infestations) | 1 (1)
Sinus Thrombosis (General disorders) | 1 (1) — Incidental finding from review of study MRI scan.
Medication Related (General disorders) | 3 (3)
Musculoskeletal Pain or Injury (Musculoskeletal and connective tissue disorders) | 4 (4)
Peripheral Vascular Disease (Vascular disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1)
Obstructive Sleep Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Syncope/Pre-Syncope (Cardiac disorders) | 1 (1)
Worsening Chronic Heart Failure (Cardiac disorders) | 9 (12)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ICD System Therapy (N=154)
MRI Incidental Finding (General disorders) | 24 (25)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators agree to submit copies of any manuscript proposed for publication to Sponsor for review at least 30 days in advance of submission for publication or presentation. Sponsor may extend such review period for another 90 days to file patent applications or take other steps to protect its intellectual property interests, or to remove from the paper or presentation any language that is detrimental to Sponsor's intellectual property interests.